CLINICAL TRIAL: NCT03821259
Title: Post-traumatic Stress Disorder (PTSD) Symptoms in Later Life: the Contribution of Cumulative Trauma Exposure, Emotion Regulation, Group Identifications, and Socioeconomic Deprivation
Brief Title: Post-traumatic Stress Disorder (PTSD) Symptoms in Later Life
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Tayside (Other Government)
Responsible Party: Sponsor
Other Study IDs: CAHSS1802/04
Record Dates: First submitted 2018-12-19; First posted 2019-01-29 (Actual); Results first posted 2020-06-23 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-06

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older adults with mental health history: Eligible participants, aged 65 and over, will be established in treatment for PTSD, anxiety or depression in the Older Adult Psychological Therapies service.
  Interventions: Other: Psychological measures

INTERVENTIONS:
Other: Psychological measures — Participants will be asked to provide basic demographic information and to complete five measures, screening for cognitive impermanent and measuring PTSD symptoms, lifetime trauma exposure, emotion regulation and group identification.

SUMMARY:
Older adults are becoming a growing proportion of people utilising mental health services. However, the needs of this population are poorly understood despite the evidence that mental health conditions are manifested differently in old age. One of those conditions is Post Traumatic Stress Disorder (PTSD) which has been associated with an increased risk of adverse outcomes in old age, including health problems, difficulties in daily functioning, less satisfaction with life and multiple psychiatric co-morbidities, such as depression and anxiety. Despite the serious consequences, PTSD symptoms in old age tend to be underreported or misperceived as a physical illness or part of an ageing process.

Traumatic life experiences do not necessarily lead to PTSD. Psychological resources, including emotional stability and social support, allow individuals to find appropriate coping strategies and maintain well-being in old age. Group identification, defined as a sense of belonging to a specific group, influences the response to social support and may be important in predicting distress in old age. On the other hand, socioeconomic deprivation is likely to increase this distress as exposure to traumatic events is more prevalent in disadvantaged populations.

The present study will investigate the impact of those factors on PTSD symptoms in later life. The researcher will recruit 85 older adults from the Older People Psychological Therapies Service, who are in receipt of psychological treatment for PTSD, anxiety or depression. Participants will be asked to provide basic demographic information, which will be used to describe the participant characteristics and to estimate the degree of socioeconomic deprivation. Participants will also complete five measures to screen for cognitive impairment and measure PTSD symptoms, lifetime trauma exposure, emotion regulation and group identification.

The findings will help improve the diagnostic process and development of psychological treatments for PTSD in older adults by expanding our knowledge of this condition in later life.

DETAILED DESCRIPTION:
Aim of the study:

To investigate the importance and relative contribution of interpersonal and intra-individual factors, including lifetime trauma exposure, emotion regulation, social group belonging and socioeconomic deprivation in predicting PTSD symptoms in older adults.

Primary research questions:

1. Will greater lifetime trauma exposure predict higher levels of PTSD symptoms in older adults?
2. Will greater difficulties in emotion regulation predict higher levels of PTSD symptoms in older adults?
3. Will a lower number of group identifications predict higher levels of PTSD symptoms in older adults?
4. Will higher levels of socioeconomic deprivation predict higher levels of PTSD symptoms in older adults?

Secondary research questions:

1. What is the relative contribution of lifetime trauma exposure in predicting levels of PTSD symptoms in older adults?
2. What is the relative contribution of difficulties in emotion regulation in predicting levels of PTSD symptoms in older adults?
3. What is the relative contribution of group identifications in predicting levels of PTSD symptoms in older adults?
4. What is the relative contribution of socioeconomic deprivation in predicting levels of PTSD symptoms in older adults?

Design:

The study will employ a cross-sectional, within-groups design. An opportunistic clinical sample of older adults, aged 65 and over, in receipt of psychological treatment for PTSD, anxiety or depression in the Older People Psychological Therapies Service in NHS Tayside will be recruited. Participants will be asked to provide basic demographic information and to complete five measures, screening for cognitive impermanent and measuring PTSD symptoms, lifetime trauma exposure, emotion regulation and group identification. Correlation and multiple regression analyses will be used to answer the research hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years and over
* In receipt of psychological treatment for PTSD, anxiety or depression
* Fluent English speaker
* Ability to give consent

Exclusion Criteria:

* Cognitive impairment (MoCA ≤20)
* Under investigation for or a confirmed diagnosis of dementia
* Currently experiencing an episode of a serious mental illness, e.g. psychosis
* Ongoing substance misuse
* Ongoing serious risk issues (i.e. risk of harm to self and others, suicidality)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: An opportunistic clinical sample of older adults, aged 65 and over, in receipt of psychological treatment for PTSD, anxiety or depression in the Older People Psychological Therapies Service in NHS Tayside will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klaudia Suchorab, MSc, Principal Investigator — NHS Tayside/University of Edinburgh
Locations (1):
- Tayside Older People Psychological Therapies service, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study recruited an opportunistic sample of suitable participants who were identified and initially approached about the study by a psychologist involved in their care. Consequently no participants were excluded following their enrolment in the study.
Groups:
- Older Adults With Mental Health History: Eligible participants, aged 65 and over in receipt of psychological treatment for PTSD, anxiety or depression, were recruited within the Older Adult Psychological Therapies service.
Period: Overall Study
Arm/Group | Older Adults With Mental Health History
Started | 88
Completed | 88
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Older Adults With Mental Health History
Number analyzed (Participants) | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.17 (4.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 88
The Civilian Version of the PTSD Checklist (PCL-C) [Mean (Standard Deviation); unit: units on a scale] — The Civilian Version of the PTSD Checklist (PCL-C; Blanchard, Jones-Alexander, Buckley, & Forneris, 1996; Weathers, Litz, Herman, Huska, & Keane, 1993) measures PTSD symptoms in the civilian population. Participants answered 17 items by rating levels of distress caused by each symptom in the past month on a 5-point scale (1 = not at all to 5 = extremely). Total scores range from 17 to 85. Higher scores indicate greater symptom severity.
  units on a scale | 42.14 (14.47)

OUTCOME MEASURES:

1. Primary Outcome: The Trauma History Questionnaire (THQ; Green, 1996)
Description: This questionnaire measures lifetime exposure to a range of potentially traumatic experiences in three broad areas of (1) crime-related events, (2) general trauma and disasters, as well as (3) unwanted sexual experiences and physical violence, and (4) other unspecified extraordinarily stressful event . Participants will be required to answer 24 items in a yes/no. Total scores range from 0 to 24. Scores for subscales are as following: (1) crime-related events: 0 - 4; (2) general trauma and disasters: 0 - 13; (3) unwanted sexual experiences and physical violence: 0 - 6; (4) other: 0 -1. Higher scores indicate more traumatic events. The THQ was developed to be applicable to various populations and has been widely used in research. In a recent review of studies employing this measure, the THQ demonstrated sound psychometric properties, including a good interrater reliability and construct validity.
Time Frame: through study completion, an average of 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Older Adults With Mental Health History: Eligible participants, aged 65 and over in receipt of psychological treatment for anxiety or depression, were recruited within the Older Adult Psychological Therapies service.
Arm/Group | Older Adults With Mental Health History
Number analyzed (Participants) | 88
score on a scale
  Total number of traumatic events | 5.93 (3.42)
  Crime-related events | 0.76 (0.88)
  General trauma and disasters | 3.81 (2.09)
  Unwanted sexual experiences and physical violence | 0.97 (1.37)

2. Primary Outcome: The Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004)
Description: This questionnaire measures six aspects of emotion regulation, including (1) acceptance of emotional responses, (2) engagement in goal-directed behaviours, (3) impulse control, (4) emotional awareness, (5) access to emotion regulation strategies and (6) emotional clarity. Participants will be required to answer 36 items by indicating the frequency of each item on a 5-point scale ranging from 1='almost never' to 5='almost always'. The total score ranges from 36 to 180. Subscales will be explored for the purpose of this study. The score ranges for each subscale are as following: (1) acceptance of emotional responses: 6 - 30, (2) engagement in goal-directed behaviours: 5 - 25, (3) impulse control: 6 - 30, (4) emotional awareness: 6 - 30, (5) access to emotion regulation strategies: 8 - 40 and (6) emotional clarity: 5 - 25. Higher scores indicate greater difficulties in emotion regulation. The DERS demonstrated a good internal consistency (α=.80-.89) and acceptable validity.
Time Frame: through study completion, an average of 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Older Adults With Mental Health History
Number analyzed (Participants) | 87
score on a scale
  DERS total score | 93.63 (24.33)
  Acceptance of emotional responses | 17.20 (6.99)
  Engagement in goal-directed behaviours | 16.59 (4.76)
  Impulse control | 12.26 (5.37)
  Emotional awareness | 14.56 (4.37)
  Access to emotion regulation strategies | 21.51 (7.13)
  Emotional clarity | 11.51 (4.18)

3. Primary Outcome: The Civilian Version of the PTSD Checklist (PCL-C; Weathers, Litz, Huska & Keane, 1994)
Description: This questionnaire measures PTSD symptoms in the civilian population. Participants will be required to answer 17 items by rating the intensity of their symptoms on a 5-point scale ranging from 1='not at all' to 5='extremely'. Total scores range from 17 to 85. Higher scores indicate greater symptom severity. The PCL-C demonstrated a high internal consistency (α=.87-.94), good test-retest reliability and positive correlations with other widely used PTSD scales. It has been reported that this measure is suitable for use with older adults with a recommended cut-off score of 37 to reliably diagnose PTSD in this population.
Time Frame: through study completion, an average of 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Older Adults With Mental Health History
Number analyzed (Participants) | 88
score on a scale | 42.14 (14.47)

4. Primary Outcome: The Group Identification Scale (GIS; Sani et al., 2012)
Description: This questionnaire measures identification with three groups (i.e. family, community and a social group chosen by the participant from the list provided, e.g. a group of friends, a voluntary group or a sports group). Identification with each group is measured with 4 items which encompass a general sense of belonging and commonality with in-group members, e.g. "I have a sense of belonging to [my group]". Participants rate their answers on a 7-point scale from 1='strongly disagree' to 7='strongly agree'. Total scores for 4 items measuring identification with each group range from 4 to 28. The cut-off score for group identification is 20, hence individuals whose total score is ≥20 across 4 items will be considered as identifying with the given group. The total number of groups the participant can identify with ranges between 0 and 3 groups. This number will be used in the final analysis. The GIS demonstrated a good internal reliability (α=.85-.92) and construct validity.
Time Frame: through study completion, an average of 6 months
Measure: Mean (Standard Deviation); unit: Number of groups participants identified
Arm/Group | Older Adults With Mental Health History
Number analyzed (Participants) | 88
Number of groups participants identified | 1.73 (1.04)

5. Primary Outcome: The Scottish Index of Multiple Deprivation (SIMD; Scottish Executive, 2016)
Description: The SIMD measures socioeconomic deprivation according to postcode information and is the only readily available measure of socioeconomic deprivation which covers the whole population of Scotland. For the purpose of this study, we will report the postcode information based on their assigned quintile, which ranges from 1 (most deprived) to 5 (least deprived).
Time Frame: through study completion, an average of 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Older Adults With Mental Health History
Number analyzed (Participants) | 88
units on a scale | 3.31 (1.27)

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Older Adults With Mental Health History
All-Cause Mortality (participants affected / at risk) | 0/88
Serious Adverse Events (participants affected / at risk) | 0/88
Other Adverse Events (participants affected / at risk) | 0/88

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/59/NCT03821259/Prot_SAP_000.pdf